CLINICAL TRIAL: NCT04519918
Title: Clinical Application of Artificial Oocyte Activation Technique (AOA) in Assisted Reproduction Technology
Brief Title: Clinical Application of Artificial Oocyte Activation Technique (AOA) in ART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOA
Record Dates: First submitted 2020-07-30; First posted 2020-08-20 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Fertilization
Keywords: Fertilization failure; Artificial Oocyte Activation (AOA); Calcium ionophore; Fertilization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard ICSI procedure (No Intervention): a single spermatozoon was injected into the ooplasm.
- Chemical oocyte activation (Experimental): After CaCl2 was injected, the oocytes were transferred into the calcium ionophore A23187 activation solution for two times of post-ICSI AOA.
  Interventions: Behavioral: AOA
- Mechanical oocyte activation (Experimental): Mechanical stimulation was done before standard ICSI procedure, then the oocytes were transferred into the calcium ionophore A23187 activation solution for two times of post-ICSI AOA.
  Interventions: Behavioral: AOA

INTERVENTIONS:
Behavioral: AOA — AOA represents an invasive non-physiological technique.
  Arms: Chemical oocyte activation; Mechanical oocyte activation

SUMMARY:
Oocyte activation is an imperative stage in the initiation of embryo development during the fertilization. Indeed, the entrance of sperm into the oocyte causes sequences of calcium oscillations in its cytoplasm, regulating a series of molecular events called oocyte activation. The intracytoplasmic sperm injection (ICSI) has allowed fertilization in couples with severe male factor infertility. But, there was still fertilization failure or low fertilization occurs in ICSI cycles. It has reported that insufficient of oocyte activation is the important cause of fertilization failure. Artificial oocyte activation (AOA) represents an effective technique, can restore the calcium oscillations to improve the fertilization. Here, the investigators explore the effective of different AOA methods including oocyte was injected CaCl2 or mechanical stimulated then treated with calcium ionophore.

DETAILED DESCRIPTION:
The ICSI procedure improves fertilization rates in cases of male factor infertility. However, fertilization failure still occurs in 1-5% in ICSI cycles. The main cause of failed fertilization is failure to complete oocyte activation. Oocyte activation involves a multitude of molecular changes. The investigators use a variety of mechanical, electrical, and chemical methods to trigger the calcium oscillations necessary to activate oocytes. During mechanical activation of oocytes, oolemmas are pierced using a microneedle to trigger a calcium influx. Another method for mechanical oocyte activation is the direct microinjection of calcium into the oocyte to increase intracellular calcium. It has been described with the use of calcium ionophore A23187, which can mimic the natural pattern of calcium rise. Mechanical and chemical activation are the most commonly used methods for artificial oocyte activation, can mimic calcium oscillations resulting in successful fertilization. AOA, a highly specialized fertilization technique that can be added to conventional ICSI to overcome fertilization failure in patients that had failed fertilization or poor quality embryos history.

When the number of retrieved oocytes was >10, sibling oocytes were divided into 3 groups to perform the standard ICSI procedure (control group), chemical AOA (A1 experiment group) or mechanical AOA (A2 experiment group). When the number of retrieved oocytes was 6-10, sibling oocytes were randomized 1:1 to perform the chemical AOA (A1 experiment group) or mechanical AOA (A2 experiment group). The number of retrieved oocytes was 1-5, all oocytes were perform the chemical AOA. Control group, a single spermatozoon was injected into the ooplasm, standard ICSI procedure. A1 experiment group, were treated by injecting CaCl2 concurrently with ICSI followed by sequential exposure of calcium ionophore A23187 activation solution for two times of post-ICSI AOA. A2 experiment group, mechanical stimulation was done before standard ICSI procedure, then the oocytes were transferred into the calcium ionophore A23187 activation solution for two times of post-ICSI AOA. The investigators want to establish the effective and safe of different AOA methods, to improve the fertilization outcome and embryo quality, and finally obtain healthy offspring.

ELIGIBILITY:
Inclusion Criteria:

* The patients suffered at least one complete fertilization failure or low fertilization rate after performing standard ICSI in previous cycle. Low fertilization was defined as less than 33% fertilization rate.
* The patients suffered at least 2 cycles complete fertilization failure or low fertilization rate after performing IVF in previous cycle. Low fertilization was defined as less than 33% fertilization rate.
* The sperm of the patients has the following characteristics: globozoospermia, acrosomal deletion or small, severe head deformity, etc.
* Sperm of testicular origin and/or sperm that has been freeze-thawed.
* The sperm was PLC-ζ missing.
* The MII oocytes were IVM cultured and/or freeze-thawed.
* The patients suffered at least 2 cycles no available embryos, because of the embryo development block or fragmentation.

Exclusion Criteria:

* Normal fertilization IVF/ICSI cycles.

Ages: 22 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of AOA on fertilization | 12 months
  Assess the normal fertilization rate (2PN rate)

SECONDARY OUTCOMES:
Efficacy of AOA on embryo quality | 12 months
  Assess the good-quality embryo rate
Efficacy of AOA on clinical outcome | 24 months
  Assess the live-birth rate

CONTACTS AND LOCATIONS:
Overall Officials: Li Bo, Doctor, Study Chair — Reproductive Medicine Center, Tangdu Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China